CLINICAL TRIAL: NCT01862159
Title: Risk Factors Predicting Serious Complications With Laparoscopic Gastric Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Region Örebro County (Other)
Collaborators: Scandinavian Obesity Surgery Registry (Unknown)
Responsible Party: Principal Investigator, Erik Stenberg, MD, MD, Region Örebro County
Other Study IDs: EPN 2012/039
Record Dates: First submitted 2013-05-02; First posted 2013-05-24 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-04

CONDITIONS: Postoperative Complications
Keywords: bariatric surgery; postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Operated patients: Patients undergoing laparoscopic gastric bypass surgery between 1st of May 2007 until 30th of september 2012
  Interventions: Procedure: laparoscopic gastric bypass surgery

INTERVENTIONS:
Procedure: laparoscopic gastric bypass surgery — laparoscopic gastric bypass surgery

SUMMARY:
The rate of serious complications are relatively low in bariatric surgery today, but still 3-4 % will suffer from a serious complication. There are factors known before the surgery or during the operation that are likely to increase the risk for a serious complication. If the investigators are aware of these we can optimize the patients risk factors prior to the operation or at least increase the awareness of the increased risk in some patients given the presence of risk factors.

DETAILED DESCRIPTION:
Data is collected prospectively to the Scandinavian Obesity Surgery Registry. Today all 44 clinics performing bariatric surgery in Sweden submits data on baseline characteristics, operational data and data from a 30 days, 1 year, 2 years and 5 years follow up for all patients. The database is compared annually to the Swedish civil registry to cover all mortality.

From the database we will identify patients who underwent a bariatric procedure between May 1st 2007 and September 30th 2012. Patients undergoing other bariatric procedures than laparoscopic gastric bypass or revisional surgery will be excluded.

The data will be analyzed with "Chi-2" test, logarithmic regression, linear regression or t-test when appropriate. Odds ratio will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Undergoing laparoscopic gastric bypass surgery and included in the Scandinavian Obesity Surgery Registry

Exclusion Criteria:

Undergoing other bariatric procedure than laparoscopic gastric bypass. Revisional surgery is excluded.

Lost to follow up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing bariatric surgery in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 25038 (Actual)
Dates: Start 2007-05; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingmar Näslund, MD, PhD, Study Chair — The Scandinavian Obesity Surgery Registry; Erik Stenberg, MD, Principal Investigator — Region Örebro County
Locations (1):
- University Hospital Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Scandinavian Obesity Surgery Registry — http://www.ucr.uu.se/soreg/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Operated Patients
Started | 25038
Completed | 25038
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Operated Patients: All patients operated with a laparoscopic gastric bypass procedure in Sweden during the inclusion period.
Arm/Group | Operated Patients
Number analyzed (Participants) | 25038
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19017
  Male | 6021
Region of Enrollment [Number; unit: participants]
  Sweden | 25038

OUTCOME MEASURES:

1. Primary Outcome: Serious Complications
Description: Graded as Clavien 3b or more (for patients entered in the registry after January 1st 2010)
Time Frame: 30 days or the postoperative hospital stay if longer than 30 days
Population: All patients operated after Jan 1, 2010
Measure: Count of Participants; unit: Participants
Arm/Group | Operated Patients
Number analyzed (Participants) | 18737
Participants | 630

2. Secondary Outcome: Operating Time
Description: length of the operation
Time Frame: operation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Operated Patients
Number analyzed (Participants) | 25038
minutes | 77.2 (38.10)

3. Secondary Outcome: Length of Stay
Description: Length of stay after the primary operation
Time Frame: 30 days or the postoperative hospital stay if longer than 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Operated Patients
Number analyzed (Participants) | 25038
days | 2.3 (3.17)

4. Secondary Outcome: Specific Postoperative Complications
Description: Any complication (Anastomotic leakage/abscesses, bleeding, small bowel obstruction, stomal ulcera, cardiovascular complications, pulmonary complications, venous thromboembolism, port site complication, other complication)
Time Frame: 30 days or the postoperative hospital stay if longer than 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Operated Patients
Number analyzed (Participants) | 25038
Participants | 2180

ADVERSE EVENTS:
Arm/Group | Operated Patients
All-Cause Mortality (participants affected / at risk) | 11/25038
Serious Adverse Events (participants affected / at risk) | 630/18737
Other Adverse Events (participants affected / at risk) | 2180/25038
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operated Patients (N=18737)
Serious adverse event (Gastrointestinal disorders) | 630 (630) — Any postoperative complication resulting in intervention under general anesthesia, organ failure or mortality (that is Clavien-Dindo 3b or more)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operated Patients (N=25038)
Any postoperative complication (Gastrointestinal disorders) | 2180 (2180) — Any deviation from a normal postoperative course (that is Clavien-Dindo grade 1 or more)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No